CLINICAL TRIAL: NCT04012177
Title: Nutritional Support and Prophylaxis Doses of Azithromycin for Pregnant Women to Improve Birth Outcomes in the Peri-urban Slums of Karachi, Pakistan -a Randomized Controlled Trial
Brief Title: Nutritional Support and Prophylaxis Doses of Azithromycin for Pregnant Women - Mumta Pregnant Women Trial
Acronym: MumtaPW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vital Pakistan Trust (Other)
Collaborators: Aga Khan University (Other)
Responsible Party: Principal Investigator, Yasir Shafiq, Senior Manager, Research and Programs, Vital Pakistan Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 004-VPT-IRB-18
Record Dates: First submitted 2019-07-01; First posted 2019-07-09 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Undernutrition
MeSH Terms: conditions — Malnutrition | interventions — Azithromycin; Choline; Niacinamide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Arm (No Intervention): Arm-A: Standard antenatal care (ANC) counseling, service provision and nutrition counseling (World Health Organization (WHO) standard)
- Nutrition only Arm (Experimental): Arm-B:Balanced-energy protein (BEP), ready-to-use utrition supplement for at least 6 months + Standard ANC counseling, service provision and nutrition counseling (WHO standard)
  Interventions: Dietary Supplement: Balanced-energy protein (BEP)
- Nutrition plus Azithromycin Arm (Experimental): Arm-C:Balanced-energy protein (BEP), ready-to-use nutrition supplement for at least 6 months + 2000 mg of Azithromycin at week 20 and 28 of pregnancy + Standard ANC counseling, service provision and nutrition counseling (WHO standard).
  Interventions: Dietary Supplement: Balanced-energy protein (BEP); Drug: Azithromycin Tablets
- Nutrition plus Choline and Nicotinamide Arm (Experimental): Arm-D: Balanced-energy protein (BEP), ready-to-use nutrition supplement for at least 6 months + Choline 450 and Nicotinamide 100 mg (1 each once daily orally starting from week 20 until birth outcome) + Standard ANC counseling, service provision and nutrition counseling (WHO standard).
  Interventions: Dietary Supplement: Balanced-energy protein (BEP); Drug: Azithromycin Tablets; Drug: Choline Bitartrate; Drug: Nicotinamide

INTERVENTIONS:
Dietary Supplement: Balanced-energy protein (BEP) — Pregnant women in the intervention arms will receive approximately 800 Kcal/day and around 16-21 gram of protein in a day in the form of ready-to-use supplement.
  Other Names: Ready-to-use-supplementary food (RUSF)
  Arms: Nutrition only Arm; Nutrition plus Azithromycin Arm; Nutrition plus Choline and Nicotinamide Arm
Drug: Azithromycin Tablets — Pregnant women randomized in Arm C will received two doses of 2000 mg of Azithromycin (4 tablets of 500 mg) oral at week 20 and 28 of pregnancy.
  Other Names: Zetro
  Arms: Nutrition plus Azithromycin Arm; Nutrition plus Choline and Nicotinamide Arm
Drug: Choline Bitartrate — Pregnant women randomized in Arm D will received 450 mg of Choline orally once daily, starting from week 20 weeks of pregnancy until birth outcome
  Other Names: Choline
  Arms: Nutrition plus Choline and Nicotinamide Arm
Drug: Nicotinamide — Pregnant women randomized in Arm D will received 100 mg of Nicotinamide orally once daily, starting from week 20 weeks of pregnancy until birth outcome
  Arms: Nutrition plus Choline and Nicotinamide Arm

SUMMARY:
This four arm trial envisions to generate robust evidence for use of a fortified balanced energy-protein supplement to pregnant women for at least 6 months, alone versus in combination of Azithromycin (AZM) prophylaxis (two prophylaxis oral doses) versus in combination with both AZM prophylaxis (two prophylaxis oral doses) plus oral Choline and Nicotinamide supplementation; to see the impact on birth weight and length of newborn soon after birth (approximately within 72 hours). This is an open label, community-based, randomized controlled trial in peri-urban settings of Karachi, Pakistan, where the outcome assessor will be blinded. The comparison groups are control arm (only routine ANC care and nutritional counseling), nutrition only arm, nutrition plus AZM arm, and nutrition plus Choline and Nicotinamide arm.

DETAILED DESCRIPTION:
Maternal under nutrition has a critical role in etiology of poor perinatal outcomes like low birth weight (LBW), accounting for 60-80% of all neonatal deaths and impacting nearly 20 million newborns overall. In Pakistan, nearly half of the households are food insecure with or without hunger. Great disparities exist between urban-rural and within urban disadvantaged populations living in the poorest of slums. In Sindh province alone, 72% of households are food insecure and 50% are with moderate to severe hunger. Around 18% of the married woman of reproductive age in Pakistan, are underweight and deficient of different micronutrients for example, 42% and 41% of women are Vitamin A and Zinc deficient, respectively.. This impacts childhood stunting, wasting, and underweight, prevalence of which, among under-five children is around 44%, 15% and 31%, respectively in Pakistan. WHO antenatal care (ANC) guidelines recommend the use of fortified balanced energy-protein supplements during pregnancy, but there is a lack of guidance on the best product/supplement for use in a particular setting. Until recently, the WHO ANC guidelines has made no recommendations on the use of these supplements in food insecure and undernourished settings. This is an area that required further research. Additionally, there is emerging literature on use of Choline and Nicotinamide during pregnancy and its potential additional impact on birth outcomes including growth and development after prenatal supplementation with Choline and Nicotinamide.

Apart from nutrition supplement, the prophylaxis use of antibiotics, especially AZM is also under strong debate, as many studies have shown improvements in birth outcomes in low middle income settings. The possible mechanism of AZM may be explained through reduction in the risk of maternal infections during pregnancy. A systematic review showed that prophylaxis may reduce the risk of postpartum endometritis, preterm rupture of membranes and gonococcal infection when given routinely to all pregnant women With no effect on birth outcome but there were several biases reported such as high loss to follow-ups and limited numbers of included studies.. Therefore, robust evidence is needed via a field trial in the local context to evaluate the efficacy and effectiveness of the locally-produced, balanced energy-protein supplement alone or in combination with prophylaxis dose of AZM or balanced energy-protein supplement alone or in combination with Choline and Nicotinamide to pregnant woman on maternal and birth outcomes in low-income and food insecure settings. This could help to draw inferences for larger public health policy-making. This investment is specifically aiming to look at what impact a newly formulated nutritional supplement for pregnant and lactating women (PLW) can have on improving birth outcomes and as well as its potential to reduce wasting, stunting and underweight in infants.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between ≥8 and < 19 weeks confirmed by ultrasound
* Able to give written voluntary informed consent.
* Permanent resident within the surveillance area, i.e. woman should be resident of the area for last 6 months at least to be considered as part of surveillance.
* Willing to spend the whole pregnancy duration after registration in trial within surveillance area until the birth outcome.
* Singleton and viable fetus on ultrasound
* Not working woman, and available for ANC and compliance visits at home.
* Previously not enrolled in pregnant woman trial.
* Previously not enrolled in Lactating woman trials.

Exclusion Criteria:

* Having Mid-upper-arm-circumference of pregnant of ≥30.5 cm
* Having known food allergies if reported by woman (like peanut, lentils)

Ages: 13 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1884 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Birth weight of newborn | To be assessed within 72 hours of birth
  Weight of the newborn assess in gram to assess the difference among four arms

SECONDARY OUTCOMES:
Birth length of newborn | To be assessed within 72 hours of birth
  Length of the newborn assess in cm to assess the difference among four arms

OTHER OUTCOMES:
Maternal hemoglobin | At enrollment and 32 weeks of pregnancy
  Assessed in (gm/dl) through Hemocue for all who are agree to assess the difference among four arms
Maternal Ferritin level | At enrollment and 32 weeks of pregnancy
  To assess the difference among four arms (ng/ml)
Maternal Vitamin D level | At enrolment and 32 weeks of pregnancy
  To assess the difference among four arms (ng/ml)
Cord blood | At birth
  Sub-sample - 50 live births in each arm to assess the difference in term of micro- and macro-nutrients and antibodies status.
Plasma for proteomic analysis | At week 19 and 32 of pregnancy
  Sub-sample - 50 women in each arm to gain in-depth analysis of proteome which potentially impact (if any) by administration of Azithromycin
Plasma for Niacin metabolites | At enrolment and 32 weeks of pregnancy
  Sub-sample - 50 women in each arm to assess the comparison among difference arm to see how these level of metabolites are different among four arm compared to those who received extra daily dose.
Urine for Choline metabolites | At enrolment and 32 weeks of pregnancy
  Sub-sample - 50 women in each arm to see how these level of metabolites are different among four arm compared to those who received extra daily dose.
Magnetic resonance imaging (MRI) of infants (post birth outcomes) | 6 and 12 months of infant's age
  Sub-sample - 50 infants of mothers each arm who will have their birth outcomes to assess brain morphology and volume of infants, using portable MRI machine "Hyperfine".
Global Scale for Early Development assessment | 6 and 12 months of infant's age
  Sub-sample - 250 infants of mothers each arm who will have their birth outcomes to assess child neurodevelopment progress, using Global Scale for Early Development (GSED)' tool. Mean scores will be compared between the arms; better scores will predict optimal neurodevelopment according to age.
Mullen assessment | 6 and 12 months of infant's age
  Sub-sample - 250 infants of mothers each arm who will have their birth outcomes to assess child neurodevelopment progress, using 'Mullen' tool. Mean scores will be compared between the arms; better scores will predict optimal neurodevelopment according to age.
Hammersmith Neurological Examinations | 6 and 12 months of infant's age
  Sub-sample - 250 infants of mothers each arm who will have their birth outcomes to assess child neurodevelopment progress, using 'Hammersmith Neurological Examinations (HINE)' tool. Mean scores will be compared between the arms; better scores will predict optimal neurodevelopment according to age.
Maternal depression | At week 19 and 32 of pregnancy and then at 6 and 12 month post-partum
  Maternal depression will be assessed using Patient Health Questionnaire (PHQ-9) during antenatal period and postnatal period. Depression scarring will be comparing scoring between the arm. Further, we will assess and compare depression severity (in any) from 'None minimal' (0-4 score) to 'Severe' (20-27 score)
Maternal and infant stool microbiome | At week 19 and 32 of pregnancy for mother, and then at 1-2, 3-4 and 5-6 and 12 months post-partum for mother-infant dyad
  Sub-sample - 50 women and the infant in each arm to assess and compared for stool microbiome
Maternal and infant stool Lipocalin-2 | At week 19 and 32 of pregnancy for mother, and then at 1-2, 3-4 and 5-6 and 12 months post-partum for mother-infant dyad
  Sub-sample - 50 women and the infant in each arm to assess and compared Lipocalin-2 (ng/gm)
Maternal and infant stool Carlprotectin | At week 19 and 32 of pregnancy for mother, and then at 1-2, 3-4 and 5-6 and 12 months post-partum for mother-infant dyad
  Sub-sample - 50 women and the infant in each arm to assess and compared Carlprotectin (ug/gm)
Maternal and infant stool Myeloperoxidase (MPO) | At week 19 and 32 of pregnancy for mother, and then at 1-2, 3-4 and 5-6 and 12 months post-partum for mother-infant dyad
  Sub-sample - 50 women and the infant in each arm to assess and compared Myeloperoxidase (ng/ml*dilution factor)
Maternal and infant stool TaqMan assay | At week 19 and 32 of pregnancy for mother, and then at 1-2, 3-4 and 5-6 and 12 months post-partum for mother-infant dyad
  Sub-sample - 50 women and the infant in each arm to assess and compared different colonies
Maternal and infant stool Bifido species | At week 19 and 32 of pregnancy for mother, and then at 1-2, 3-4 and 5-6 and 12 months post-partum for mother-infant dyad
  Sub-sample - 50 women and the infant in each arm to assess and compared for Bifido species
Metabolomic work - Maternal during pregnancy | At enrolment and 32 week of pregnancy
  All women who are agreed in each arm, for metabolomic work using 'Volumetric Absorptive Microsampling (VAM)
Metabolomic work - Mother-Infant dyad | 1-2, 3-4 and 5-6 and 12 months post-partum for mother-infant dyad
  Sub-sample - 50 women and the infant in each arm for metabolomic work using 'Volumetric Absorptive Microsampling (VAM) Infants - sub-sample of 50 infants of same enrolled women in each arm for metabolomic work using'Volumetric Absorptive Microsampling (VAM)
Human milk oligosaccharides | within 72 hours of birth
  Sub-sample - 50 women in each arm to assess and compare breastmilk oligosaccharides
Breastmilk quality | within 72 hours of birth
  Sub-sample - 50 women in each arm to assess and compare breastmilk quality (macro-and micro-nutrients)
Breastmilk microbiome | within 72 hours of birth
  Sub-sample - 50 women in each arm to assess and compare microbiomes.
Breastmilk immunoglobulin | within 72 hours of birth
  Sub-sample - 50 women in each arm to assess immunoglobulins in the breastmilk

CONTACTS AND LOCATIONS:
Overall Officials: Yasir Shafiq, MSc, Principal Investigator — Vital Pakistan Trust; Ameer Muhammad, MSc, Principal Investigator — Vital Pakistan Trust; Fyezah Jehan, MSc, Principal Investigator — Aga Khan University; Muhammad Imran Nisar, MSc, Principal Investigator — Aga Khan University
Locations (1):
- Peri-urban slum (Rehri Goth), Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muhammad A, Fazal ZZ, Baloch B, Nisar I, Jehan F, Shafiq Y. Nutritional support and prophylaxis of azithromycin for pregnant women to improve birth outcomes in peri-urban slums of Karachi, Pakistan-a protocol of multi-arm assessor-blinded randomized controlled trial (Mumta PW trial). Trials. 2022 Jan 3;23(1):2. doi: 10.1186/s13063-021-05960-9. PMID 34980232